CLINICAL TRIAL: NCT04488510
Title: Pathogens Involved in Secondary Infections During Severe Forms of Covid-19 Pneumonia: COVAP Study
Brief Title: Pathogens Involved in Secondary Infections During Severe Forms of Covid-19 Pneumonia:
Acronym: COVAP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Centre Hospitalier Victor Dupouy (Other)
Responsible Party: Sponsor
Other Study IDs: COVAP
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Ventilator Associated Pneumonia; Nosocomial Pneumonia
Keywords: Pneumonia under mechanical ventilation; ICU; covid19; coronavirus; nosocomial pneumonia; bacteria
MeSH Terms: conditions — COVID-19; Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During the inclusion, a 4 ml citrate tube of blood in addition to the usual management assessment and aspiration of tracheal secretions will be performed at D1, D3 and D7. Tracheal aspiration is performed systematically in order to limit patient congestion and the risk of atelectasis.

SUMMARY:
A Respiratory infection with the SARS-CoV2 virus is associated with a major risk of viral pneumonia that can lead to respiratory distress requiring resuscitation. In the most severe forms, it may require mechanical ventilation or even lead to an acute respiratory distress syndrome with a particularly poor prognosis. The SARS-CoV2 is a single-stranded RNA virus of positive polarity and belongs to the beta genus of Coronaviruses. SARS-CoV2 is responsible for the third epidemic in less than twenty years secondary to a Coronavirus (SARS-CoV then MERS-CoV) and if the mortality associated with it is lower than that of previous strains, notably MERS-CoV, its spread is considerably big. As a result, the number of patients developing respiratory distress requiring invasive mechanical ventilation is high, with prolonged ventilation duration in these situations

DETAILED DESCRIPTION:
Patients requiring invasive mechanical ventilation are at risk of secondary, nosocomial, a hospitalization in the ICU service and can affect up to 40% of ventilated patients. The occurrence of ventilator-associated pneumonia is associated with an increase in the duration of mechanical ventilation and its effect on mortality remains uncertain under general conditions. The mechanisms underlying the occurrence of lower respiratory infection during invasive mechanical ventilation are numerous, depending for the most part on two distinct elements: the occurrence of transcolonisation, which will secondarily promote colonisation of the lower respiratory tract, and the modification of the competence of the immune system in its response to aggression by microbial agents whose pathogenicity is highly variable.

Throughout the infection by SARS-CoV2, the theoretical risk of secondary respiratory infection during mechanical ventilation is important due to the intrication of three concomitant phenomena: direct pulmonary aggression, which will alter the functionality of local immunity, the "cytokinic storm", responsible for the severity of the respiratory picture that motivated intubation and the need for mechanical ventilation leading inevitably to transcolonisation. Despite all of these pathophysiological arguments, very little data are available on the possibility of secondary low respiratory tract infection occurring during SARS-CoV2 infection and more generally during Coronarivus infections. even though all of these elements are well known and widely studied, very little data are currently available on the potential interaction between Coronaviruses and bacteria. The importance of this issue is very significant as recent observations tend to show a relative rarity of the occurrence of secondary lung infections during mechanical ventilation and the population of smokers, subject to chronic obstructive bronchitis (usually particularly susceptible to bacterial superinfections), does not appear to be more affected than that of non-smokers although the current data are very partial.

The research is prospective, non interventional study that involves patients suffering from another severe form a COVID-19 infection: the nosocomial pneumonia under mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years old
* French-speaking patient
* Patient whose COVID-19 infection was diagnosed by either a laboratory test, PCR or any other commercial or public health test.
* Adult acute respiratory distress syndrome according to the Berlin definition
* Pneumonia acquired under mechanical ventilation defined according to the criteria of international companies

Exclusion Criteria:

* Patient/family or proxy opposing participation in the study
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under the safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged over 18 years, infected by the COVID-19 with a severe form of pneumonia especially the nosocomial pneumonia acquired under mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Research of the bacteria responsible for nosocomial pneumonia | 6 months
  Establishing a biobank of the bacterial agents responsible for nosocomial pneumonia acquired under mechanical ventilation in order to: better understand the particularities of the bacteria responsible and obtain the "clinical" strains for in vitro studies that will be carried out secondarily.

SECONDARY OUTCOMES:
Additional evaluations to the study | 6 months
  Evaluation of the adhesion properties to the bronchial epithelium (LPS peculiarities of Gram-negative bacteria, the interaction with the virus in in vitro models and the different molecules of interest in the collected bronchial secretions).

CONTACTS AND LOCATIONS:
Overall Officials: François PHILLIPART, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France